CLINICAL TRIAL: NCT04237779
Title: The Effects of Intratesticular PRP Injection
Brief Title: The Effects of Intratesticular PRP Injection in Men With Azoospermia or Cryptozoospermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Bulent Tiras, Prof., Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATADEK 2019-4/23
Record Dates: First submitted 2020-01-12; First posted 2020-01-23 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Azoospermia, Nonobstructive
MeSH Terms: conditions — Azoospermia, Nonobstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection into at least one testis (Experimental): Autologous blood obtained from peripheral vein will be used to prepare PRP following standard protocols. PRP injection will be performed under local anesthesia. Sperm analysis, testicular volumes (using orchiometer), serum FSH and testosterone measurements will be re-evaluated at 8 weeks post-procedure. On the third month after the procedure, presence of spermatozoa will be reassessed in microTESE material.
  Interventions: Biological: PRP injection into at least one testis

INTERVENTIONS:
Biological: PRP injection into at least one testis — Autologous blood obtained from peripheral vein will be used to prepare PRP following standard protocols. PRP injection will be performed under local anesthesia. Sperm analysis, testicular volumes (using orchiometer), serum FSH and testosterone measurements will be re-evaluated at 8 weeks post-procedure. On the third month after the procedure, presence of spermatozoa will be reassessed in micro testicular sperm extraction (TESE) material.

SUMMARY:
The study will be conducted in men with a diagnosis of non-obstructive azoospermia or cryptozoospermia after obtaining written informed consent. The diagnosis of azoospermia and cryptozoospermia will be based on two semen analyses performed at least 15 days apart, followed by a documented micro testicular sperm extraction (TESE). A detailed history will be obtained, physical examination and laboratory evaluation will be performed prior to treatment. In physical examination, testicular volumes will be evaluated using an orchiometer. Serum FSH and testosterone values will be determined. PRP will be prepared by centrifugation of approximately 20 ml autologous blood obtained by phlebotomy. PRP (3 ml) will be administered into the seminiferous tubule or interstitial space of each testis. Sperm analysis, testicular volume (using orchiometer), serum FSH and testosterone levels will be reevaluated at 8 weeks post-procedure. Micro TESE will performed on the third month after PRP procedure.

DETAILED DESCRIPTION:
Platelet-rich plasma (PRP) is a unique autologous agent derived from blood that is rich in growth factors, cytokines, and hormones; it has been reported to reduce oxidative stress and reactive oxygen species generation and upregulate the expression of various antioxidant enzymes. PRP is used in a variety of clinical applications in cell therapy. Based on World Health Organization guidelines, azoospermia is diagnosed when the absence of sperm is observed in two semen samples. Based on World Health Organization (WHO), cryptozoospermia is diagnosed when spermatozoa cannot be observed in a fresh semen sample; however, it is found after an extended centrifugation and microscopic search. All patients require a clinical work-up with physical examination, endocrine evaluation (follicle stimulating hormone (FSH), luteinizing hormone (LH) and testosterone) and genetic analysis. Scrotal and transrectal ultrasounds will be performed as indicated. Platelet-rich plasma (PRP), with its rich growth factor composition, has proven beneficial in regenerative therapy. The potential therapeutic role of PRP has not been studied in testis for non-obstructive azoospermia and cryptozoospermia. The investigators will investigate sperm parameters in non-obstructive azoospermic and crypotozoospermic patients treated with PRP.

ELIGIBILITY:
Inclusion Criteria:

* Azoospermia in at least 2 prior semen analysis.
* Diagnosis of Non-Obstructive Azoospermia or Diagnosis of Cryptozoospermia

Exclusion Criteria:

* Obstructive Azospermia
* Anatomical abnormalities in the genital tract,
* Cancer,
* Hepatitis
* Patients with systemic medical problems
* Patients with chromosomal disorders

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Azoospermia in at least 2 prior semen analysis. Diagnosis of Non-Obstructive Azoospermia or Diagnosis of Cryptozoospermia
Enrollment: 200 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
sperm formation | 6 months
  Number of participants with testicular PRP treatment as assessed by testicular sperm extraction, change from azoospermia or cryptozoospermia to presence of sperm during TESE procedure

SECONDARY OUTCOMES:
IVF outcomes | 12 months
  Number of participants with testicular PRP after TESE as assessed by number of clinical pregnancies, change in the clinical pregnancy rates with IVF treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yigit Cakiroglu, Assoc.Prof., Study Director — Acibadem University
Locations (1):
- Acıbadem Maslak Hospital IVF Unit, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhurat R, Sukesh M. Principles and Methods of Preparation of Platelet-Rich Plasma: A Review and Author's Perspective. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):189-97. doi: 10.4103/0974-2077.150734. PMID 25722595
- [Result] Dehghani F, Sotoude N, Bordbar H, Panjeshahin MR, Karbalay-Doust S. The use of platelet-rich plasma (PRP) to improve structural impairment of rat testis induced by busulfan. Platelets. 2019;30(4):513-520. doi: 10.1080/09537104.2018.1478400. Epub 2018 Jun 8. PMID 29883240